CLINICAL TRIAL: NCT05776433
Title: The Effects of Extremity With Lymphedema on Posture, Upper Extremity Functions, and Quality of Life in Patients With Lymphedema After Unilateral Breast Cancer
Brief Title: The Effects of Upper Extremity Lymphedema on Posture, Upper Extremity Functions, and Quality of Life
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Simla Turan, Principal Investigator, Yeditepe University
Other Study IDs: YU-FTR-ST-01
Record Dates: First submitted 2023-02-22; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer Related Lymphedema; Breast Cancer-Related Arm Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Unilateral upper extremity lymphedema women after breast cancer treatment: The study group consisted of women aged 18-50 years with unilateral upper extremity lymphedema after breast cancer treatment.

SUMMARY:
This study aims to examine the effects of lymphedema extremity on upper extremity function, posture and quality of life in patients who develop upper extremity lymphedema after unilateral breast cancer. Twenty-seven volunteers (27Female) diagnosed with upper extremity lymphedema after unilateral breast cancer treatment by a specialist physician between May 2022 and October 2022 were included in the study. Upper extremity circumference measurements of the individuals were performed on the healthy and affected sides. A goniometer measured both sides' upper extremity range of motion (ROM). The New York Posture Analysis (NYPA) was used for posture evaluation. Upper extremity functions were assessed by the Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire and the Lymphedema Functionality, Disability and Health Questionnaire (Lymph-ICF). Quality of life was assessed by Upper Extremity Lymphedema-27 (ULL-27) and Quality of Life Measure for Limb Lymphedema -Arm (LYMQOL- Arm).

DETAILED DESCRIPTION:
This study aims to examine the effects of lymphedema extremity on upper extremity function, posture and quality of life in patients who develop upper extremity lymphedema after unilateral breast cancer. Twenty-seven volunteers (27Female) diagnosed with upper extremity lymphedema after unilateral breast cancer treatment by a specialist physician between May 2022 and October 2022 were included in the study. Upper extremity circumference measurements of the individuals were performed on the healthy and affected sides. A goniometer measured both sides' upper extremity range of motion (ROM). The New York Posture Analysis (NYPA) was used for posture evaluation. Upper extremity functions were assessed by the Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire and the Lymphedema Functionality, Disability and Health Questionnaire (Lymph-ICF). Quality of life was assessed by Upper Extremity Lymphedema-27 (ULL-27) and Quality of Life Measure for Limb Lymphedema -Arm (LYMQOL- Arm).

The hypotheses of our study:

Hypothesis 0 (H0):

There is no relationship between upper extremity function, posture and quality of life in patients with upper extremity lymphedema after unilateral breast cancer treatment.

Hypothesis 1 (H1):

There is a relationship between upper extremity function, posture and quality of life in patients with upper extremity lymphedema after unilateral breast cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Be between the ages of 18-50
* Having had unilateral breast cancer
* At least one year since breast cancer treatment
* No active metastases

Exclusion Criteria:

* Arthritis
* Fibromyalgia syndrome
* Neurological diseases
* Mental illnesses
* Myopathic diseases
* Bilateral upper extremity lymphedema
* Inability to communicate and cooperate
* Presence of any orthopaedic disease in the affected upper extremity
* Having scoliosis
* Having cognitive problems

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 27 female
Study Population: The sample of the study consists of patients who applied to Istanbul Dr Nazif Bağrıaçık Kadıköy Hospital in Istanbul between May 2022 and October 2022 and were diagnosed with upper extremity lymphedema after unilateral breast cancer by the doctor.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand (DASH) | 10 minutes
  It is a disability/symptom scoring system based on a self-report system of 30 items developed to evaluate upper extremity-specific physical functions and symptoms. The DASH questionnaire, which consists of three parts, contains 30 questions. Of these, 21 questions evaluate the patient's difficulty during physical activity, five assess symptoms (pain, activity-related pain, tingling, weakness, difficulty in movement), and the remaining four evaluate the patient's social function, work, sleep, and self-confidence. Questions are scored from 1 to 5 (1: no difficulty, 2: mild difficulty, 3: medium difficulty, 4: extreme difficulty, 5: none at all). The total score is between 0-100. The DASH score is calculated using the formula [sum of answers/n-1] x 25 (n=number of questions answered).
Lymphedema Functionality, Disability, and Health Questionnaire (Lymph-ICF) | 10 minutes
  Lymph-ICF, a descriptive and evaluation tool, consists of 29 questions about the functional impairments, activity limitations, and participation restrictions reported by patients with breast cancer-related lymphedema. Physical function, mental function, home activities, mobility activities, and life and social activities are the five main components into which the questionnaire is subdivided. There is a visual analogue scale next to each question, and the patient marks the answer that suits themself. While calculating the survey score, the score of each subsection is found by summing and dividing by the number of questions answered. The total score is obtained by adding the scores of the subsections. A high score indicates that the effect on the quality of life is high.
Upper Extremity Lymphedema-27 (ULL-27) | 10 minutes
  ULL-27 is a quality-of-life questionnaire evaluating upper extremity lymphedema as three components. The scale deals with physical, psychological and social components and consists of 27 questions. A 5-point Likert score (1=strongly disagree, 5=strongly agree) is used in the scale. The first 15 questions evaluate the physical component, questions between 16-22 evaluate the psychological component, and questions between 23-27 evaluate the social component. The lowest score is 27, and the highest score is 135. A high score on the scale indicates that lymphedema negatively affects the quality of life. The physical score consists of a total of fifteen questions, and this score of the person is between min 15 and 75. The psychological score consists of seven questions, with a minimum of 7 and a maximum of 35 points. There are five questions for the social score, with a minimum of 5 and a maximum of 25 points.
Quality of Life Measure for Limb Lymphedema-Arm (LYMQOL-Arm) | 10 minutes
  The LYMQOL-Arm, primarily as a self-assessment report questionnaire assessing the symptoms of lymphedema in the upper extremity and the ability to perform functional activities in patients with breast cancer-associated lymphedema. There are five subsections in the 21-question survey. These are upper extremity function (questions 1a-h,2,3), appearance (questions 4-8), symptoms (questions 9-14), emotional state (questions 15-20), and general quality of life ( 21st question). In the first 20 questions, there are four options for each question: none (1 point), a little (2 points), quite (3 points), and a lot (4 points). The scores of these subsections are summed up within themselves and divided by the number of questions answered. In the 21st question, the patient is asked to give a value between 0 and 10 for the quality of life. High scores for the first 20 questions and low scores for the 21st question indicate poor quality of life.
The New York Posture Analysis (NYPA) | 5 minutes
  Posture is the optimal form of all body parts about the whole body and the adjacent segment. This assessment test evaluates posture disorders that occur in 13 different body regions. The scoring of the test is as follows; A score of 5 is given if the person has a proper posture, 3 points if there is a moderate impairment, and 1 point if there is a severe disorder. The maximum score obtained at the end of the test is 65, and the minimum is 13. The standard evaluation criteria developed for the test are as follows for the total score; >=45: very good, 40-44: good, 30-39: medium, 20-29: weak, <=19:bad

OTHER OUTCOMES:
Upper Extremity Circumference Measurement | 1 hour
  Circumference measurements were evaluated for both upper extremities. Markings were made every 4 cm, assuming the wrist pivot point. Upper extremity circumference measurements were made at 4 cm intervals up to the axilla. The difference between the affected and healthy sides was determined.
Goniometric Measurements | 1 hour
  The active range of motion (ROM) of both shoulders (affected and healthy) was measured with a goniometer. Flexion and abduction were measured in the supine position and extension in the prone position. Internal and external rotations were measured in the supine position with the shoulder 90° abducted and the elbow 90° flexion. A difference of ≥20° between the affected and unaffected sides was considered a limitation in the ROM of the affected side.

CONTACTS AND LOCATIONS:
Overall Officials: Simla Turan, Principal Investigator — Yeditepe University; Feryal Subaşı, Study Director — Yeditepe University
Locations (1):
- Dr. Nazif Bağrıaçık Kadıköy Hospital, Kadıköy, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] DiSipio T, Rye S, Newman B, Hayes S. Incidence of unilateral arm lymphoedema after breast cancer: a systematic review and meta-analysis. Lancet Oncol. 2013 May;14(6):500-15. doi: 10.1016/S1470-2045(13)70076-7. Epub 2013 Mar 27. PMID 23540561
- [Result] Ahmed RL, Prizment A, Lazovich D, Schmitz KH, Folsom AR. Lymphedema and quality of life in breast cancer survivors: the Iowa Women's Health Study. J Clin Oncol. 2008 Dec 10;26(35):5689-96. doi: 10.1200/JCO.2008.16.4731. Epub 2008 Nov 10. PMID 19001331
- [Result] Taghian NR, Miller CL, Jammallo LS, O'Toole J, Skolny MN. Lymphedema following breast cancer treatment and impact on quality of life: a review. Crit Rev Oncol Hematol. 2014 Dec;92(3):227-34. doi: 10.1016/j.critrevonc.2014.06.004. Epub 2014 Jul 2. PMID 25085806
- [Result] Haddad CA, Saad M, Perez Mdel C, Miranda Junior F. Assessment of posture and joint movements of the upper limbs of patients after mastectomy and lymphadenectomy. Einstein (Sao Paulo). 2013 Dec;11(4):426-34. doi: 10.1590/s1679-45082013000400004. PMID 24488379
- [Result] Leray H, Malloizel-Delaunay J, Lusque A, Chantalat E, Bouglon L, Chollet C, Chaput B, Garmy-Susini B, Yannoutsos A, Vaysse C. Body Mass Index as a Major Risk Factor for Severe Breast Cancer-Related Lymphedema. Lymphat Res Biol. 2020 Dec;18(6):510-516. doi: 10.1089/lrb.2019.0009. Epub 2020 Apr 13. PMID 32283042
- [Result] Ridner SH, Dietrich MS, Stewart BR, Armer JM. Body mass index and breast cancer treatment-related lymphedema. Support Care Cancer. 2011 Jun;19(6):853-7. doi: 10.1007/s00520-011-1089-9. Epub 2011 Jan 16. PMID 21240649
- [Result] Belmonte R, Messaggi-Sartor M, Ferrer M, Pont A, Escalada F. Prospective study of shoulder strength, shoulder range of motion, and lymphedema in breast cancer patients from pre-surgery to 5 years after ALND or SLNB. Support Care Cancer. 2018 Sep;26(9):3277-3287. doi: 10.1007/s00520-018-4186-1. Epub 2018 Apr 12. PMID 29651594
- [Result] Levangie PK, Drouin J. Magnitude of late effects of breast cancer treatments on shoulder function: a systematic review. Breast Cancer Res Treat. 2009 Jul;116(1):1-15. doi: 10.1007/s10549-008-0246-4. Epub 2008 Nov 25. PMID 19031114
- [Result] Babasaheb SS, Rajesh KK, Yeshwant KS, Patil S. Analysis of Spinal Dysfunction in Breast Cancer Survivors with Lymphedema. Asian Pac J Cancer Prev. 2021 Jun 1;22(6):1869-1873. doi: 10.31557/APJCP.2021.22.6.1869. PMID 34181345
- [Result] Dawes DJ, Meterissian S, Goldberg M, Mayo NE. Impact of lymphoedema on arm function and health-related quality of life in women following breast cancer surgery. J Rehabil Med. 2008 Aug;40(8):651-8. doi: 10.2340/16501977-0232. PMID 19020699
- [Result] Park JE, Jang HJ, Seo KS. Quality of life, upper extremity function and the effect of lymphedema treatment in breast cancer related lymphedema patients. Ann Rehabil Med. 2012 Apr;36(2):240-7. doi: 10.5535/arm.2012.36.2.240. Epub 2012 Apr 30. PMID 22639749
- [Result] Pusic AL, Cemal Y, Albornoz C, Klassen A, Cano S, Sulimanoff I, Hernandez M, Massey M, Cordeiro P, Morrow M, Mehrara B. Quality of life among breast cancer patients with lymphedema: a systematic review of patient-reported outcome instruments and outcomes. J Cancer Surviv. 2013 Mar;7(1):83-92. doi: 10.1007/s11764-012-0247-5. Epub 2012 Dec 5. PMID 23212603
- [Result] Rietman JS, Dijkstra PU, Hoekstra HJ, Eisma WH, Szabo BG, Groothoff JW, Geertzen JH. Late morbidity after treatment of breast cancer in relation to daily activities and quality of life: a systematic review. Eur J Surg Oncol. 2003 Apr;29(3):229-38. doi: 10.1053/ejso.2002.1403. PMID 12657232
- [Result] Ridner SH, Bonner CM, Deng J, Sinclair VG. Voices from the shadows: living with lymphedema. Cancer Nurs. 2012 Jan-Feb;35(1):E18-26. doi: 10.1097/NCC.0b013e31821404c0. PMID 21558848